CLINICAL TRIAL: NCT04727229
Title: Stellate Ganglion Block for Major Depressive Disorder: A Randomized Controlled Pilot Trial
Brief Title: Stellate Ganglion Block for Major Depressive Disorder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-301
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
Keywords: Feasibility trial; Stellate Ganglion Block; Bupivacaine
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine Hydrochloride (Experimental): Injection of Bupivacaine Hydrochloride 0.5% near the stellate ganglion.
  Interventions: Drug: Bupivacaine Hydrochloride
- Normal Saline Solution (Placebo Comparator): Injection of Normal Saline near the stellate ganglion
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Injection of Bupivacaine near the stellate ganglion
  Arms: Bupivacaine Hydrochloride
Drug: Normal Saline — Injection of Normal Saline near the stellate ganglion
  Arms: Normal Saline Solution

SUMMARY:
This is a feasibility study, to investigate a new treatment option for major depressive disorders by performing a Stellate Ganglion Block (SGB). A SGB is an injection of local anesthetic into the sympathetic nervous system (peripheral nervous system) located in the lower part of the neck, to relieve pain in the head, neck, upper arm, and upper chest.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 65 years of age
2. Major depressive disorder without psychotic symptoms according to DSM-5 criteria
3. Hamilton Depression Rating Scale (HAMD)>17
4. Current major depressive episode as confirmed by the Mini International Neuropsychiatric Interview (MINI)
5. Failure of at least two trials of antidepressant therapy during the current episode
6. Capacity to provide informed consent

Exclusion Criteria:

1. Depression secondary to stroke, cancer or other severe medical illness
2. Major Depressive Episode in people with Bipolar Disorder.
3. Dementia
4. Post-Traumatic Stress Disorder (PTSD)
5. Acute suicidality defined as score ≥3 on HAMD item 3
6. Previous electroconvulsive therapy
7. Known history of intolerance of hypersensitivity to local anesthetic
8. Current substance abuse or dependence (except for caffeine or nicotine dependence) and/or recent history (last 12 months) of current alcohol abuse or dependence, as defined in DSM-5 criteria
9. Unwilling to maintain current antidepressant regimen.
10. A clinical finding/condition that is unstable or that, in the opinion of the investigator(s) would negatively be affected by an SGB (e.g. movement disorder where patient is unable to lie still for injection or anatomical variants making an SGB impractical).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Feasibility, Recruitment, Acceptability, Safety, | 1 year
  Recruitment rate, withdrawal rate, adherence rate, frequency of adverse events

SECONDARY OUTCOMES:
Change in the symptoms of depression | 6 weeks
  ≥ 50% reduction in the Montgomery-Åsberg Depression Rating Scale (MADRS) score. The MADRS score range from 0 to 6 = no depression; from 7 to 19 = mild depression, 20 to 34 = moderate depression, 35 and greater = severe depression, and a total score of 60 or greater = very severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Karim Ladha, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data has been planned to be shared with other researchers at this point since this is a feasibility study with only 10 participants.

REFERENCES:
- [Result] Sussman D, Tassone VK, Gholamali Nezhad F, Wu M, Adamsahib F, Mattina GF, Pazmino-Canizares J, Demchenko I, Jung H, Lou W, Ladha KS, Bhat V. Local Injection for Treating Mood Disorders (LIFT-MOOD): A Pilot Feasibility RCT of Stellate Ganglion Block for Treatment-Resistant Depression. Chronic Stress (Thousand Oaks). 2023 Mar 3;7:24705470231160315. doi: 10.1177/24705470231160315. eCollection 2023 Jan-Dec. PMID 36895443